CLINICAL TRIAL: NCT02389985
Title: A Phase Ib/II Study of CRLX101 in Combination With Weekly Paclitaxel in Patients With Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: A Study of CRLX101(NLG207) in Combination With Weekly Paclitaxel in Patients With Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRLX101-209
Record Dates: First submitted 2015-03-02; First posted 2015-03-17 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — IT-101; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRLX101 and weekly paclitaxel (Experimental): CRLX101 and weekly paclitaxel administered by IV on days 1 and 15 of a 28 day cycle. Paclitaxel only is administered by IV on day 8.
  Interventions: Drug: CRLX101; Drug: Paclitaxel

INTERVENTIONS:
Drug: CRLX101
  Other Names: NLG207
Drug: Paclitaxel
  Other Names: Taxol

SUMMARY:
The purpose of this study is to estimate the maximum tolerated doses (MTD) of CRLX101 when administered in combination with weekly paclitaxel in women with recurrent or persistent, epithelial ovarian, fallopian tube or primary peritoneal cancer.

Determine through pharmacokinetic evaluation(sometimes described as what the body does to a drug, refers to the movement of drug into, through and out of the body-the time and course of its absorption, bioavailability, distribution, metabolism, and excretion) whether or not the disposition of paclitaxel is affected by the concurrent administration of CRLX101.

DETAILED DESCRIPTION:
Recurrent ovarian cancer represents a therapeutic challenge. Patients with resistant disease, showing progression within six months of platinum-containing therapy, have a poor prognosis, with median overall survival (OS) approximately 12 months.Ultimately most patients with recurrent disease ultimately develop platinum resistance, and novel strategies are needed.

In this setting the most active agents are pegylated liposomal doxorubicin (PLD), paclitaxel and topotecan. Multiple trials have demonstrated that combination therapy produces increased toxicity without improved efficacy.

This study proposes to examine the combination of CRLX101 in combination with weekly paclitaxel. Preclinical studies show synergistic activity in the SKOV3 human ovarian cancer xenograft ovarian cancer cell lines (14), as well as in vivo (15,16), perhaps via an antiangiogenic mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. Histologic documentation of the original primary tumor is required via the pathology report.
2. Patient must have measurable disease or detectable (non-measurable) disease:

   Measurable disease will be defined by RECIST 1.1.
3. Patients must have adequate bone marrow, renal, hepatic, and neurologic functions
4. Patients should be free of active infection requiring parenteral antibiotics.
5. Any other prior therapy directed at the malignant tumor, including chemotherapy, bevacizumab or other biologic or targeted agents and immunologic agents, must be discontinued at least 21 days (three weeks) prior to registration.
6. Any prior radiation therapy must be discontinued at least four weeks prior to registration.
7. Major surgery within 28 days (four weeks) prior to registration.
8. Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease.
9. Patients must have a GOG performance status of 0 or 1.
10. Patients who will be enrolled under protocol amendment # 2 must have previously received bevacizumab, either discontinued due to intolerability, or progressed after at least 2 cycles of bevacizumab

Exclusion Criteria:

1. Patients who have had previous treatment with:

   * CRLX101 or with any topoisomerase I therapy;
   * Weekly paclitaxel for recurrent or persistent disease.
2. Patients with a history of other invasive malignancies, with the exception of non-melanoma skin, are excluded if:

   * There is any evidence of other malignancy being present within the last three years;
   * Previous cancer treatment contraindicates this protocol therapy.
3. Patients with known active hepatitis or HIV.
4. Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first dose of study drug.
5. Patients with clinically significant cardiovascular disease.
6. Patients with serous non-healing wound, ulcer, or bone fracture.
7. Patients with active bleeding or pathologic conditions that carry high risk of bleeding
8. Patients with clinical symptoms or signs of gastrointestinal obstruction and who require parenteral hydration and/or nutrition.
9. Patients with active infection requiring parenteral antibiotics.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2018-06-04 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
1. To estimate the maximum tolerated doses (MTD) of CRLX101 when administered in combination with weekly paclitaxel in women with recurrent or persistent, epithelial ovarian, fallopian tube or primary peritoneal cancer. | 6 months
  The highest dose with <2 patients with DLTs out of 6 DLT-evaluable patients

SECONDARY OUTCOMES:
Comparison of pharmacokinetic perimeters including max concentration (Cmax), time to maximum concentration (Tmax), AUC, elimination half-life for CRLX101 and paclitaxel | 6 months
  PK

OTHER OUTCOMES:
2. To assess the overall safety and tolerability of CRLX101 in combination with weekly paclitaxel. | 6 months
  AEs, changes in clinical status, vital signs, and laboratory data
To assess the anti-tumor activity of CRLX101 when administered concomitantly with weekly paclitaxel in patients with recurrent or persistent epithelial ovarian fallopian tube or primary peritoneal cancer. | 6 months
  PFS per RECIST 1.1 with scans every 2 cycles

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma / Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Derived] Duska LR, Krasner CN, O'Malley DM, Hays JL, Modesitt SC, Mathews CA, Moore KN, Thaker PH, Miller A, Purdy C, Zamboni WC, Lucas AT, Supko JG, Schilder RJ. A phase Ib/II and pharmacokinetic study of EP0057 (formerly CRLX101) in combination with weekly paclitaxel in patients with recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal cancer. Gynecol Oncol. 2021 Mar;160(3):688-695. doi: 10.1016/j.ygyno.2020.12.025. Epub 2020 Dec 31. PMID 33390325